CLINICAL TRIAL: NCT07166315
Title: Clinical Characteristics, Treatment Patterns and Outcomes in Patients With axSpA and PsA Following Initiation of Bimekizumab, Risankizumab, Guselkumab, Upadacitinib or a TNF Inhibitor
Brief Title: Treatment Effectiveness in People With axSpA or PsA Starting Treatment With Bimekizumab, Risankizumab, Guselkumab, Upadacitinib, or a TNF Inhibitor
Status: Recruiting | Type: Observational
Sponsor: Adelphi Real World (Industry)
Responsible Party: Sponsor
Other Study IDs: AG9827
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Axial Spondylarthritis (axSpA); Psoriatic Arthritis (PsA)
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Axial spondyloarthritis (axSpA): Patients diagnosed with axial spondyloarthritis (axSpA) who are initiating treatment with bimekizumab, upadacitinib, or a tumour necrosis factor-alpha inhibitor.
  Interventions: Other: observational study
- Psoriatic arthritis (PsA): Patients diagnosed with psoriatic arthritis (PsA) who are initiating treatment with bimekizumab, upadacitinib, risankizumab, guselkumab or a tumour necrosis factor-alpha inhibitor.
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — This is an observational study based on existing treatments prescribed prior to inclusion. No interventions are given as part of this research.

SUMMARY:
This observational study will target patients with axial spondyloarthritis (axSpA) and psoriatic arthritis (PsA) who have started treatment with bimekizumab, upadacitinib, risankizumab, guselkumab, or a tumour necrosis factor-alpha inhibitor (e.g., adalimumab or etanercept) at NHS hospitals in the United Kingdom. Information from patients' medical records will be collected, and patients will complete surveys about their experiences with their treatment. The study will look at treatment effectiveness from both healthcare professionals' and patients' points of view.

DETAILED DESCRIPTION:
Patient experience surveys will be administered prospectively throughout the study period, whereas the review of patients' medical records will be conducted retrospectively towards the end of the study period.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a clinical diagnosis of axial spondyloarthritis (axSpA) or psoriatic arthritis (PsA).
* Participant has been prescribed advanced therapy within one month prior to enrolment in the study, to treat their axSpA or PsA.
* Participant is aged 18 years or older at enrolment.

Exclusion Criteria:

-Participation in a clinical trial at enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from patients attending NHS hospitals and related healthcare sites targeted across the United Kingdom, including England, Scotland, Wales, and Northern Ireland. These sites are secondary and tertiary care centres where patients with axial spondyloarthritis or psoriatic arthritis are routinely managed by rheumatology services.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants that have achieved Low Disease Activity (LDA) at 12 months. | At 12 months
Number of participants that have achieved Minimal Disease Activity (MDA) at 12 months. | At 12 months
Change from baseline in PROM scores at 12 months. | At 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Royal National Hospital for Rheumatic Diseases, Bath, Somerset, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) from this study will not be shared with other researchers. In accordance with the study protocol and relevant data protection regulations, including GDPR, only aggregated data and summary results will be made available for scientific dissemination. All data provided will be fully anonymized and presented in aggregate form to ensure participant confidentiality and privacy. No individual-level data or information that could identify participants will be shared outside of the authorized study team.